CLINICAL TRIAL: NCT03310554
Title: Prevention of Duodenobiliary Reflux Via Suspended Overlength Biliary Stents in Patients With Biliary Stricture
Brief Title: Suspended Overlength Biliary Stents Preventing Duodenobiliary Reflux in Patients With Biliary Stricture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Huang Yonghui, Chief physician, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: M2017187
Record Dates: First submitted 2017-10-11; First posted 2017-10-16 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Bile Duct Stricture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinding of endoscopists and patients is impossible.But the endoscopists are not involved in the assessment of outcomes. The outcomes assessments are performed by reviewing physicians blinded to the randomization process. The data manager and statistician are not blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 26cm suspended overlength biliary stents group (Experimental)
  Interventions: Procedure: 26cm suspended overlength biliary stents
- 30cm suspended overlength biliary stents group (Experimental)
  Interventions: Procedure: 30cm suspended overlength biliary stents
- ordinary plastic biliary stents group (Other)
  Interventions: Procedure: ordinary plastic biliary stents

INTERVENTIONS:
Procedure: 26cm suspended overlength biliary stents — The test group will be placed 26cm suspended overlength biliary stents in introhepatic bile duct in ERCP
  Arms: 26cm suspended overlength biliary stents group
Procedure: 30cm suspended overlength biliary stents — The test group will be placed 30cm suspended overlength biliary stents in introhepatic bile duct in ERCP
  Arms: 30cm suspended overlength biliary stents group
Procedure: ordinary plastic biliary stents — The control group will be placed ordinary plastic biliary stents in bile duct in ERCP
  Arms: ordinary plastic biliary stents group

SUMMARY:
Endoscopic insertion of plastic or metal stents in bile duct under endoscopic retrograde cholangiopancreatography is a well established treatment of distal malignant biliary obstruction.Biliary stents are widely used to relieve symptoms of malignant biliary stricture.Now, the mainly used biliary stents include plastic and metal stents. The main limitation of long time plastic stents is stents occlusion. Biliary plastic stents are changed every 2 to 3 months due to an expected median patency from 77 to 126 days.Metal stents present a lower risk of recurring biliary occlusion, yet high cost and stents occlusion are eventually inevitable. The mechanism of biliary stents occlusion include biliary sluge of the accumulation of bacteria and duodenal biliary reflux .The anti-reflux barrier of Oddi's sphincter disappears after the insertion of biliary stents and the presure in bile duct lowers the duodenals, which cause the retrograde flow of duodenal material into the biliary ducts. Besides, ordinary biliary plastic stent is short which can also shortens the length of duodenal biliary reflux . Therefore, trying to prevent the duodenal biliary reflux is very important in reducing biliary stents occlusion and it is gradually concerned by clinical researchers. Some studies have showed that plastic stents with antireflux valves can effectively reduce the biliary stent stricture and prolong the stents patency, which means reducing duodenobiliary reflux is surely useful for keeping biliary stent patency.So,we assume to explore an innovatively suspended overlength biliary stents (made from nasobiliary tube with length of 26cm or 30cm) as substitution for ordinary biliary plastic stent to prevent the duodenobiliary reflux by extending the length of duodenal content reflux and avoid the stents shift via suspending in intrahepatic duct. In this study,we will design a randomized controlled trial to compare the patency of different length of suspended overlength biliary stents and ordinary plastic biliary stents in patients with distal malignant biliary obstruction to evaluate the effect and safety of suspended overlength biliary stents for the prevention of duodenobiliary reflux and the effect of different length of the stents.

DETAILED DESCRIPTION:
Endoscopic insertion of plastic or metal stents in bile duct under endoscopic retrograde cholangiopancreatography is a well established treatment of distal malignant biliary obstruction.Biliary stents are widely used to relieve symptoms of malignant biliary stricture.Now, the mainly used biliary stents include plastic and metal stents. The main limitation of long time plastic stents is stents occlusion. Biliary plastic stents are changed every 2 to 3 months due to an expected median patency from 77 to 126 days.Metal stents present a lower risk of recurring biliary occlusion, yet high cost and stents occlusion are eventually inevitable. The mechanism of biliary stents occlusion include biliary sluge of the accumulation of bacteria and duodenal biliary reflux .The anti-reflux barrier of Oddi's sphincter disappears after the insertion of biliary stents and the presure in bile duct lowers the duodenals, which cause the retrograde flow of duodenal material into the biliary ducts. Besides, ordinary biliary plastic stent is short which can also shortens the length of duodenal biliary reflux . Therefore, trying to prevent the duodenal biliary reflux is very important in reducing biliary stents occlusion and it is gradually concerned by clinical researchers. Some studies have showed that plastic stents with antireflux valves can effectively reduce the biliary stent stricture and prolong the stents patency, which means reducing duodenobiliary reflux is surely useful for keeping biliary stent patency .So,we assume to explore an innovatively suspended overlength biliary stents (made from nasobiliary tube with length of 26cm or 30cm) as substitution for ordinary biliary plastic stent to prevent the duodenobiliary reflux by extending the length of duodenal content reflux and avoid the stents shift via suspending in intrahepatic duct. In this study,we will design a randomized controlled trial to compare the patency of different length of suspended overlength biliary stents and ordinary plastic biliary stents in patients with distal malignant biliary obstruction to evaluate the effect and safety of suspended overlength biliary stents for the prevention of duodenobiliary reflux and the effect of different length of the stents.

The investigators will recruit patients according to admission criteria and exclusion criteria. Eligible patients with distal malignant biliary obstruction will be randomly divided into 26cm suspended overlength biliary stents group (experimental group) 、30cm suspended overlength biliary stents group (experimental group) and ordinary plastic biliary stents group (control group).The test groups will be placed the 26cm or 30cm suspended overlength biliary stents in introhepatic bile duct in ERCP. The control group will be placed ordinary plastic biliary stents in ERCP. The primary endpoint is the duration of stent patency and the rate of stent occlusion.The secondary outcomes include the mortality of each group, adverse events and the rate of technical success.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable extrahepatic malignant biliary stricture,available for insertion of biliary stents in ERCP to alleviate biliary stricture.

Exclusion Criteria:

1. Patients agree with metal biliary stents;
2. Patients with biliary stricture need double or multiple stents inserted;
3. Patients with previous surgical drainage procedure;
4. Patients with resectable biliary occlusion;
5. A guidewire could not be passed through the stricture;
6. Patients with duodenal obstruction and duodenal endoscopy could not be reached to papillary.;
7. Patients with any contraindication to endoscopic procedures or refuse informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2018-01-11 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
stent patency and stent occlusion rate | 12 months after ERCP
  Patients with symptoms of cholangitis and worsening liver function tests suggestive of cholestasis are considered as premature stent occlusion.

SECONDARY OUTCOMES:
mortality of each group | 12 months after ERCP
  We will compare the mortality of each group after the insertion of biliary stents.
adverse events | 12 months after ERCP
  Adverse events include complications of post ERCP such as pancreatitis,biliary infection, bleeding, perforation and stent migration etc.
the rate of technical success | 12 months after ERCP
  Technical success is defined as successful insertion of the stent into the bile duct during ERCP.

CONTACTS AND LOCATIONS:
Overall Officials: Yonghui Huang, archiater, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dumonceau JM, Tringali A, Blero D, Deviere J, Laugiers R, Heresbach D, Costamagna G; European Society of Gastrointestinal Endoscopy. Biliary stenting: indications, choice of stents and results: European Society of Gastrointestinal Endoscopy (ESGE) clinical guideline. Endoscopy. 2012 Mar;44(3):277-98. doi: 10.1055/s-0031-1291633. Epub 2012 Feb 1. PMID 22297801
- [Result] Libby ED, Leung JW. Prevention of biliary stent clogging: a clinical review. Am J Gastroenterol. 1996 Jul;91(7):1301-8. PMID 8677983
- [Result] Pedersen FM, Lassen AT, Schaffalitzky de Muckadell OB. Randomized trial of stent placed above and across the sphincter of Oddi in malignant bile duct obstruction. Gastrointest Endosc. 1998 Dec;48(6):574-9. doi: 10.1016/s0016-5107(98)70038-0. PMID 9852446
- [Result] van Berkel AM, Boland C, Redekop WK, Bergman JJ, Groen AK, Tytgat GN, Huibregtse K. A prospective randomized trial of Teflon versus polyethylene stents for distal malignant biliary obstruction. Endoscopy. 1998 Oct;30(8):681-6. doi: 10.1055/s-2007-1001388. PMID 9865556
- [Result] van Berkel AM, Bruno MJ, Bergman JJ, van Deventer SJ, Tytgat GN, Huibregtse K. A prospective randomized study of hydrophilic polymer-coated polyurethane versus polyethylene stents in distal malignant biliary obstruction. Endoscopy. 2003 Jun;35(6):478-82. doi: 10.1055/s-2003-39666. PMID 12783344
- [Result] Reddy DN, Banerjee R, Choung OW. Antireflux biliary stents: are they the solution to stent occlusions? Curr Gastroenterol Rep. 2006 Apr;8(2):156-60. doi: 10.1007/s11894-006-0012-x. PMID 16533479
- [Result] van Berkel AM, van Marle J, van Veen H, Groen AK, Huibregtse K. A scanning electron microscopic study of biliary stent materials. Gastrointest Endosc. 2000 Jan;51(1):19-22. doi: 10.1016/s0016-5107(00)70380-4. PMID 10625789
- [Result] Soehendra N, Reynders-Frederix V. Palliative bile duct drainage - a new endoscopic method of introducing a transpapillary drain. Endoscopy. 1980 Jan;12(1):8-11. doi: 10.1055/s-2007-1021702. PMID 7353562
- [Result] Wagh MS, de Bellis M, Fogel EL, Frakes JT, Johanson JF, Qaseem T, Howell DA, Lehman GA, Sherman S. Multicenter Randomized Trial of 10-French versus 11.5-French Plastic Stents for Malignant Biliary Obstruction. Diagn Ther Endosc. 2013;2013:891915. doi: 10.1155/2013/891915. Epub 2013 May 2. PMID 23737656
- [Result] Groen AK, Out T, Huibregtse K, Delzenne B, Hoek FJ, Tytgat GN. Characterization of the content of occluded biliary endoprostheses. Endoscopy. 1987 Mar;19(2):57-9. doi: 10.1055/s-2007-1018235. PMID 3106022
- [Result] Speer AG, Cotton PB, Rode J, Seddon AM, Neal CR, Holton J, Costerton JW. Biliary stent blockage with bacterial biofilm. A light and electron microscopy study. Ann Intern Med. 1988 Apr;108(4):546-53. doi: 10.7326/0003-4819-108-4-546. PMID 2450501
- [Result] Leung JW, Ling TK, Kung JL, Vallance-Owen J. The role of bacteria in the blockage of biliary stents. Gastrointest Endosc. 1988 Jan-Feb;34(1):19-22. doi: 10.1016/s0016-5107(88)71223-7. PMID 3280393
- [Result] Liu YF, Saccone GT, Thune A, Baker RA, Harvey JR, Toouli J. Sphincter of Oddi regulates flow by acting as a variable resistor to flow. Am J Physiol. 1992 Nov;263(5 Pt 1):G683-9. doi: 10.1152/ajpgi.1992.263.5.G683. PMID 1443142
- [Result] Sung JY, Leung JW, Shaffer EA, Lam K, Olson ME, Costerton JW. Ascending infection of the biliary tract after surgical sphincterotomy and biliary stenting. J Gastroenterol Hepatol. 1992 May-Jun;7(3):240-5. doi: 10.1111/j.1440-1746.1992.tb00971.x. PMID 1611012
- [Result] Donelli G, Guaglianone E, Di Rosa R, Fiocca F, Basoli A. Plastic biliary stent occlusion: factors involved and possible preventive approaches. Clin Med Res. 2007 Mar;5(1):53-60. doi: 10.3121/cmr.2007.683. PMID 17456835
- [Result] van Berkel AM, van Marle J, Groen AK, Bruno MJ. Mechanisms of biliary stent clogging: confocal laser scanning and scanning electron microscopy. Endoscopy. 2005 Aug;37(8):729-34. doi: 10.1055/s-2005-870131. PMID 16032491
- [Result] Dua KS, Reddy ND, Rao VG, Banerjee R, Medda B, Lang I. Impact of reducing duodenobiliary reflux on biliary stent patency: an in vitro evaluation and a prospective randomized clinical trial that used a biliary stent with an antireflux valve. Gastrointest Endosc. 2007 May;65(6):819-28. doi: 10.1016/j.gie.2006.09.011. Epub 2007 Mar 26. PMID 17383650
- [Result] Vihervaara H, Gronroos JM, Hurme S, Gullichsen R, Salminen P. Antireflux Versus Conventional Plastic Stent in Malignant Biliary Obstruction: A Prospective Randomized Study. J Laparoendosc Adv Surg Tech A. 2017 Jan;27(1):53-57. doi: 10.1089/lap.2016.0178. Epub 2016 Oct 18. PMID 27754790
- [Result] Rees EN, Tebbs SE, Elliott TS. Role of antimicrobial-impregnated polymer and Teflon in the prevention of biliary stent blockage. J Hosp Infect. 1998 Aug;39(4):323-9. doi: 10.1016/s0195-6701(98)90298-5. PMID 9749404
- [Result] Yang F, Ren Z, Chai Q, Cui G, Jiang L, Chen H, Feng Z, Chen X, Ji J, Zhou L, Wang W, Zheng S. A novel biliary stent coated with silver nanoparticles prolongs the unobstructed period and survival via anti-bacterial activity. Sci Rep. 2016 Feb 17;6:21714. doi: 10.1038/srep21714. PMID 26883081
- [Result] Kenawy el-R, Abdel-Hay FI, el-Raheem A, el-Shanshoury R, el-Newehy MH. Biologically active polymers: synthesis and antimicrobial activity of modified glycidyl methacrylate polymers having a quaternary ammonium and phosphonium groups. J Control Release. 1998 Jan 2;50(1-3):145-52. doi: 10.1016/s0168-3659(97)00126-0. PMID 9685881